CLINICAL TRIAL: NCT06111287
Title: : Outcomes of Trasversus Abdominis Release for Complex Abdominal Wall Hernia Repair: an Italian Multicenter Cohort Study
Brief Title: Outcomes of Trasversus Abdominis Release for Complex Abdominal Wall Hernia
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Azienda Sanitaria Locale Napoli 2 Nord (Other)
Responsible Party: Principal Investigator, Francesco Pizza, MD,PhD, Responsible for the Bariatric and Metabolic Surgery unit, Azienda Sanitaria Locale Napoli 2 Nord
Other Study IDs: 1988
Record Dates: First submitted 2023-10-23; First posted 2023-11-01 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Hernia, Abdominal; Hernia Incisional
MeSH Terms: conditions — Hernia, Abdominal; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter retrospective study analyzed data from 308 patients who underwent open Posterior Component separation with Trasversus release for primary or recurrent complex abdominal hernias between 2015 and 2020. The primary endpoint was the rate of Hernia Recurrence and Mesh Bulging at 3, 6, 12, 24, and 36 months. Secondary outcomes included surgical site events and were assessed using the Pain scale.

DETAILED DESCRIPTION:
Study design This study is reported according to the STROBE statement for cohort studies A retrospective multicentric study was conducted to analyze the surgical outcomes of patients undergoing open with Posterior Component separation with Trasversus release for inisional hernia. It was conducted according to the ethical principles stated in the Declaration of Helsinki. Written informed consent was obtained from all subjects.

Study setting and study population From January 2015 and May 2020, all the patients affected by primary or recurrent complex abdominal hernias undergoing open Posterior Component separation with Trasversus release referring to 6 centers, were considered for enrollment in the study. Inclusion criteria were age ≥16 years, primary or recurrent complex abdominal hernias with more than >10 cm midline defects Exclusion criteria were follow-up data lower than 36 months, patients with a stoma for whom closure was not planned during the abdominal hernia repair

ELIGIBILITY:
Inclusion Criteria:

* age ≥16 years,
* primary or recurrent complex abdominal hernias with more than >10 cm midline defects

Exclusion Criteria:

* follow-up data lower than 36-months, patients with a stoma for whom closure was not planned during the abdominal hernia repair

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From January 2015 and May 2020, all the patients affected by primary or recurrent complex abdominal hernias undergoing open component posterior separation with trasversus abdomen release referring to 6 centres, were considered for enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 432 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2020-05 (Actual); Study Completion 2020-07 (Actual)

PRIMARY OUTCOMES:
Hernia Recurrence | 3 months
  In details, Hernia Recurrence was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Hernia Recurrence | 6 months
  In details, Hernia Recurrence was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Hernia Recurrence | 12 months
  In details, Hernia Recurrence was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Hernia Recurrence | 24 months
  In details, Hernia Recurrence was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Hernia Recurrence | 36 months
  In details, Hernia Recurrence was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Mesh Bulging | 3 months
  In details, Mesh Bulging was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Mesh Bulging | 12 months
  In details, Mesh Bulging was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Mesh Bulging | 24 months
  In details, Mesh Bulging was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
Mesh Bulging | 36 months
  In details, Mesh Bulging was clinically defined as any visible or palpable ''blowout'' in the abdominal wall. computed tomography scan evaluation was carried out by a radiologist with 10 years of gastrointestinal computed tomography scan experience.
surgical site events | 1 months
  Regarding the surgical site events, the classification of wound events was assigned according to the likelihood and degree of wound contamination at the time of the operation, as stated in the Centre for Disease Control and Prevention wound classification (superficial, deep or organ space)
Number of patients affected by Superficial surgical site infection | 1 months
  Superficial infections according to Clavien-Dindo criteria

SECONDARY OUTCOMES:
Number of patients affected by Superficial surgical site infections | Within 30 days postoperatively
  Superficial infections according to Clavien-Dindo criteria
Number of patients affected by Deep surgical site infections | Within 30 days postoperatively
  Deep surgical site infections according to Clavien-Dindo criteria
Number of patients affected by organ space infections | Within 30 days postoperatively
  Organ space infections according to Clavien-Dindo criteria
Number of patients affected by Surgical Site Occurence | Within 30 days postoperatively
  Surgical Site Occurence Reported according to the Ventral Hernia Working Group (VHWG) definitions
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 1 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 3 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 6 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 12 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 24 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Postoperative pain | Postoperative pain will be recorded according to visual analogue scale Visual Analogue Scale at 36 month.
  Postoperative pain will be recorded according to the Visual Analogue Scale (VAS). The Visual Analogue Scale (VAS) measures pain intensity. The Visual Analogue Scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Francdesco Pizza, Napoli, Naples
  - Francesco Pizza, Naples

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: july 2024